CLINICAL TRIAL: NCT00495144
Title: A Phase I, Multi-Center, Open-Label, Dose-Escalation Study of the Safety, Pharmacokinetics and Anti-Tumor Activity of TH-302 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of the Safety, Pharmacokinetics, and Anti-Tumor Activity of TH-302 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-401
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Tumors; Hypoxia
Keywords: Phase I; Advanced Solid Tumors; Hypoxia; Prodrug; Multi-Center; Open-Label; Dose-Escalation
MeSH Terms: conditions — Neoplasms; Hypoxia | interventions — TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TH-302

SUMMARY:
This is a phase I, multi-center, open-label, dose-escalation study of TH-302 in patients with advanced solid tumors. TH-302 is a hypoxia activated product designed to exploit the hypoxic nature of tumors. The study is designed to establish the safety including the maximum tolerated dose, the pharmacokinetics, and the anti-tumor activity of TH-302.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Histologically or cytologically confirmed advanced or metastatic solid malignancy
* Advanced or metastatic solid malignancy previously treated with one or more regimens of chemotherapy or for which no effective therapy is available
* Recovered from toxicities of prior therapy
* Measurable disease by RECIST criteria (at least one target lesion)
* ECOG performance status of 0 or 1
* Life expectancy of at least 3 months
* Acceptable liver function:

  * Bilirubin ≤ 1.5 times upper limit of normal
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 times upper limit of normal (ULN); if liver metastases are present, then ≤ 5 x ULN is allowed
* Acceptable renal function:

  * Serum creatinine ≤ ULN
* Acceptable hematologic status (without hematologic support):

  * ANC ≥ 1500 cells/μL
  * Platelet count ≥ 100,000/μL
  * Hemoglobin ≥ 9.0 g/dL
* Urinalysis: No clinically significant abnormalities
* Acceptable coagulation status:

  * PT ≤ 1.3 x ULN
  * PTT ≤ 1.3 x ULN
* All women of childbearing potential must have a negative serum pregnancy test and women and men subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria:

* Prior treatment with high dose chemotherapy
* Prior radiotherapy to more than 25% of the bone marrow
* New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within 6 months prior to Day 1, or unstable arrhythmia
* Seizure disorders requiring anticonvulsant therapy
* Symptomatic brain metastases (unless previously treated and well controlled for a period of ≥ 3 months)
* Severe chronic obstructive pulmonary disease with hypoxemia or in the opinion of the investigator any physiological state leading to hypoxemia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Treatment with radiation therapy, surgery, chemotherapy, targeted therapies (erlotinib, lapatinib, etc.) or hormones within 4 weeks prior to study entry (6 weeks for nitrosoureas or Mitomycin C)
* Patients who participated in an investigational drug or device study within 28 days prior to study entry
* Known infection with HIV, hepatitis B, or hepatitis C
* Patients who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation (containing solutol and/or propylene glycol)
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of TH-302 administered weekly x 3, repeated every 4 weeks in patients with advanced solid tumors

SECONDARY OUTCOMES:
To establish the pharmacokinetics of intravenously administered TH-302
To assess the anti-tumor activity of TH-302 as measured by objective response and duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, MD, Principal Investigator — SCRI Development Innovations, LLC; Glen Weiss, MD, Principal Investigator — Translational Drug Development
Locations (7):
- United States (7):
  - TGen Drug Development Services, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - St. Mary's Medical Center, San Francisco, California
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers, Dallas, Texas

REFERENCES:
- See also: Threshold Pharmaceuticals Company Website — http://www.thresholdpharm.com